CLINICAL TRIAL: NCT03499808
Title: A Phase II Study of Isatuximab (SAR650984) (NSC-795145) for Patients With Previously Treated AL Amyloidosis
Brief Title: S1702 Isatuximab in Treating Patients With Relapsed or Refractory Primary Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1702; NCI-2017-01375 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1702 (Other: SWOG); S1702 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-02

CONDITIONS: Amorphous, Eosinophilic, and Acellular Deposit; Constipation; Diarrhea; Early Satiety; Gastrointestinal Hemorrhage; Hepatomegaly; Lymphadenopathy; Macroglossia; Nausea; Primary Systemic Amyloidosis; Purpura; Recurrent Primary Amyloidosis; Refractory Primary Amyloidosis
MeSH Terms: conditions — Constipation; Diarrhea; Gastrointestinal Hemorrhage; Hepatomegaly; Lymphadenopathy; Macroglossia; Nausea; Immunoglobulin Light-chain Amyloidosis; Purpura | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (isatuximab) (Experimental): Patients receive isatuximab IV on days 1, 8, 15, and 22 of course 1 and on days 1 and 15 of subsequent courses. Treatment repeats every 28 days for 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Isatuximab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Isatuximab — Given IV
  Other Names: Hu 38SB19; SAR 650984; SAR650984
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well isatuximab works in treating patients with primary amyloidosis that has come back or does not respond to treatment. Monoclonal antibodies, such as isatuximab, may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy as measured by the confirmed overall hematologic response rate (partial response or better) of isatuximab in relapsed/refractory systemic light chain (AL) amyloidosis.

SECONDARY OBJECTIVES:

I. To evaluate toxicities in the treatment of relapsed/refractory AL amyloidosis with isatuximab.

II. To evaluate time to hematologic response. III. To evaluate duration of response. IV. To evaluate progression-free survival (PFS). V. To evaluate overall survival (OS).

TERTIARY OBJECTIVES:

I. To evaluate efficacy of isatuximab in relapsed/refractory immunoglobulin amyloid light chain (AL) amyloidosis as measured by organ specific response rates (cardiac, renal, gastrointestinal [GI], liver, soft tissue, nerve), in the subset of patients that can be evaluated for organ response.

II. To evaluate time to organ response in the subset of patients that can be evaluated for organ response.

OUTLINE:

Patients receive isatuximab intravenously (IV) on days 1, 8, 15, and 22 of course 1 and on days 1 and 15 of subsequent courses. Treatment repeats every 28 days for 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days and then every at least every 6 months for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have relapsed or refractory primary systemic AL amyloidosis, histologically-confirmed by positive Congo red stain with green by birefringence on polarized light microscopy, OR characteristic appearance by electron microscopy AND confirmatory AL amyloid typing (mass spectrometry-based proteomic analysis or immunofluorescence)
* Patient must have measurable disease within 28 days prior to registration; serum beta2 microglobulin, serum quantitative immunoglobulins (immunoglobulin [Ig]G, IgA, and IgM), serum free kappa and lambda, and serum protein electrophoresis (SPEP) with M-protein quantification must be obtained within 14 days prior to registration
* Patient must demonstrate a difference in the involved serum free light chains (kappa or lambda) versus the uninvolved serum free light chain of >= 4.5 mg/dL within 14 days prior to registration
* Patient must have objective organ involvement defined by ONE (or more) of the following; all disease for involved organs must be assessed and documented on the AL baseline tumor assessment form

  * Kidney: albuminuria greater than or equal to 500 mg per day on a 24-hour urine specimen within 35 days prior to registration, OR prior kidney biopsy (at time of diagnosis) showing amyloid deposition
  * Heart: mean left ventricular wall thickness on echocardiogram greater than or equal to 12 mm in the absence of hypertension or valvular heart disease, OR N-terminal fragment brain natriuretic protein (NT-pro) brain natriuretic peptide (BNP) greater than 332 ng/mL provided that patient does not have impaired renal function (as defined by calculated creatinine clearance less than 25 mL/min) within 14 days prior to registration, OR prior cardiac biopsy (at time of diagnosis) showing amyloid deposition with past documented or presently noted clinical symptoms and signs supportive of a diagnosis of heart failure in the absence of an alternative explanation for heart failure
  * Liver: hepatomegaly (total liver span > 15 cm) as demonstrated by computed tomography (CT) or magnetic resonance imaging (MRI) within 35 days prior to registration OR elevated alkaline phosphatase (ALP) greater than 1.5 times the upper limit of normal within 14 days prior to registration, OR prior liver biopsy (at time of diagnosis) showing amyloid deposition
  * Gastrointestinal tract: prior biopsy showing amyloid deposition AND symptoms such as GI bleeding or persistent diarrhea (> 4 loose stools/day on most days over a consecutive 28-day period)
  * Autonomic or peripheral nervous system: orthostatic blood pressure, symptoms of nausea, early satiety, diarrhea or constipation, abnormal sensory and/or motor findings on neurologic exam, or gastric atony by gastric emptying scan; Note: pulse and blood pressure must be recorded with the patient supine (lying down), and then again after at least 1 minute, but less than 3 minutes of standing; this assessment must be repeated on 2 separate occasions (at least 1 day apart; e.g. day -3 and day -1) within a 28-day screening period
  * Soft tissue: macroglossia, or soft tissue deposits (including lymphadenopathy, recurrent peri-orbital purpura, peri-articular, skin or other soft tissue) requiring therapy
* Patients must not have active symptomatic multiple myeloma, as defined by 2015 International Myeloma Working Group (IMWG) criteria (hypercalcemia, renal failure, anemia, and bone [CRAB] criteria; bone marrow plasmacytosis > 60%); kappa: lambda ratio > 100 is acceptable only if the clinical symptoms and sign are attributable only to amyloidosis and not multiple myeloma (hemoglobin [Hgb] < 8 g/dL)
* Patient must be relapsed or refractory to at least one prior line of therapy (such as: transplant, radiation, or chemotherapy)
* Patients must have completed other systemic therapy >= 14 days or investigational drug >= 28 days prior to registration, surgery (other than biopsies) >= 21 days prior to registration, and any autologous stem cell transplant (ASCT) >= 100 days prior to registration
* Patients must not have received any or supplements which have been known to have some anti-amyloidogenic effect (such as: doxycycline; curcumin; prednisone; dexamethasone; epigallocatechin gallate [EGCG]) within 14 days prior to registration
* Patients must not have any known allergies to isatuximab or other monoclonal antibody therapies
* Patients must not have received daratumumab within 56 days prior to registration nor have been refractory to daratumumab
* Patients must not be eligible for autologous stem cell transplantation
* Patients must have a complete medical history and physical exam within 14 days prior to registration
* Within 14 days prior to registration: Total bilirubin =< 2.0 x IULN (institutional upper limit of the norm) AND
* Within 14 days prior to registration: Serum glutamic-oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) and serum glutamate pyruvate transaminase (SGPT)/alanine aminotransferase (ALT) =< 4.0 x IULN
* Creatinine clearance (CrCl) >= 25 mL/min, as measured by a 24-hour urine collection or as estimated by the Cockcroft and Gault formula; the serum creatinine value used in the calculation must have been obtained within 35 days prior to registration
* Patients must have bone marrow aspirate, including fluorescence in situ hybridization (FISH) (including: del 17p; t11;14; t4;14, t14;16; and del 13q) and cytogenetic testing (normal ? XY; and all abnormalities) within 35 days prior to registration; central pathology analysis will not be required, however the local pathology report and FISH/cytogenetic data must be submitted in Medidata RAVE
* Within 14 days prior to registration: Absolute neutrophil count (ANC) >= 1,000 cells/mcl without growth factor support, AND
* Within 14 days prior to registration: Platelets >= 75,000 cells/mcl
* Patients must have hemoglobin >= 8 g/dL within 14 days prior to registration; patients may have received transfusion if greater than 7 days prior to registration
* New York Heart Association (NYHA) < class IV heart failure
* Left ventricular ejection fraction (LVEF) by echocardiogram (ECHO) >= 35% within 35 days prior to registration; and
* NT-proBNP =< 8500 ng/L within 14 days prior to registration
* Patients must have a Zubrod performance status =< 2
* Patients must not have any clinically significant uncontrolled systemic illness, including but not limited to uncontrolled, active infection requiring intravenous antibiotics, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmias, uncontrolled hypertension, or uncontrolled diabetes mellitus

  * Uncontrolled diabetes: patients who have a diagnosis of diabetes must have an glycosylated hemoglobin (HbA1C) < 7% within 14 days prior to registration; the same criterion will be used in patients with confirmed diagnosis of diabetes mellitus who have been on a stable dietary or therapeutic regimen for this condition in the last three months
  * Uncontrolled blood pressure and hypertension: all blood pressure measurements within the 14 days prior to registration must be systolic blood pressure (SBP) =< 160 and diastolic blood pressure (DBP) =< 100; an exception can be made by a healthcare provider for a patient with a single blood pressure elevation who upon rechecking has a normal blood pressure
* Females of childbearing potential must have a negative baseline pregnancy test within 14 days prior to registration; this may be either a serum or urine pregnancy test, with a sensitivity of at least 50 mIU/mL; females of childbearing potential (FCBP) must also agree: (1) to have a pregnancy test prior to the start of each treatment cycle and (2) to either commit to continued abstinence from heterosexual intercourse or to use effective contraception while receiving study drug and for at least 12 weeks after receiving the last dose of study drug; females are considered to be of ?childbearing potential? if they have had menses at any time in the preceding 24 consecutive months; in addition to routine contraceptive methods, ?effective contraception? also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, she is responsible for beginning contraceptive measures
* Patients with evidence of hepatitis B virus (HBV) are eligible provided there is minimal hepatic injury and the patient has undetectable HBV on suppressive HBV therapy; patient must be willing to maintain adherence to HBV therapy; patients with previously treated and eradicated hepatitis C virus (HCV) who have minimal hepatic injury are eligible
* Patients who are known to be human immunodeficiency virus (HIV)-positive at registration are eligible if at time of registration they meet all other protocol eligibility criteria in addition to the following:

  * Patient has undetectable HIV viral load by standard polymerase chain reaction (PCR) clinical assay
  * Patient is willing to maintain adherence to combination antiretroviral therapy
  * Patient has no history of acquired immunodeficiency syndrome (AIDS) defining condition (other than CD4 cell count < 200 mm^3)
  * Patient is otherwise likely to have a near normal lifespan if not for the presence of relapsed/refractory amyloid
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Scott, Principal Investigator — SWOG Cancer Research Network
Locations (345):
- United States (345):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Stephens Memorial Hospital, Norway, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Parker TL, Rosenthal A, Sanchorawala V, Landau HJ, Campagnaro EL, Kapoor P, Neparidze N, Girnius S, Hagen P, Scott EC, Hoering A, Durie BGM, Orlowski RZ. Isatuximab for relapsed and/or refractory AL amyloidosis: results of a prospective phase 2 trial (SWOG S1702). Blood. 2025 Nov 20;146(21):2507-2516. doi: 10.1182/blood.2024027962. PMID 40925099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 participants were enrolled of which 35 were eligible and analyzable.
Period: Overall Study
Arm/Group | Treatment (Isatuximab)
Started | 43
Completed | 19
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Isatuximab)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: Years] | 70 [40.1 to 79.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 4
Performance Status [Count of Participants; unit: Participants] — PS 0 - Fully active, able to carry on all pre-disease performance without restriction PS 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work. PS 2- Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    PS 0 | 8
    PS 1 | 25
    PS 2 | 2
Involved Light Chain [Count of Participants; unit: Participants]
  Kappa | 10
  Lambda | 23
  None | 1
  Unknown | 1
IgG (mg/dL) [Median (Full Range); unit: mg/dL] | 700 [141 to 1689]
Organ Involvement [Count of Participants; unit: Participants]
  Single Organ Involvement | 18
  Multiple Organ involvement | 17
Mayo Cardiac Biomarker Stage [Count of Participants; unit: Participants] — Stage I: all below cutoff Stage II: 1 above Stage III: 2 above Stage IV: 3 above
  cTnT ≥0.025 ng/ml NT-proBNP ≥1,800 pg/ml FLC-diff ≥18 mg/dl
  Participants
    Stage I | 7
    Stage II | 8
    Stage III | 8
    Stage IV | 1
    Unknown | 1
    Not assessed - no cardiac involvement at baseline | 10
Plasma Cells (%, Bone Marrow) [Median (Full Range); unit: % of Bone Marrow] | 6 [0 to 30]
Kidney Involvement [Count of Participants; unit: Participants]
  Yes | 14
  No | 21
Nervous System Involvement [Count of Participants; unit: Participants]
  Yes | 9
  No | 26
Liver Involvement [Count of Participants; unit: Participants]
  Yes | 1
  No | 34
Soft Tissue Involvement [Count of Participants; unit: Participants]
  Yes | 5
  No | 30
GI Tract Involvement [Count of Participants; unit: Participants]
  Yes | 2
  No | 33
Cardiac Involvement [Count of Participants; unit: Participants]
  Yes | 25
  No | 10

OUTCOME MEASURES:

1. Primary Outcome: Assess Efficacy by Confirmed Overall Hematologic Response
Description: To assess the efficacy as measured by the confirmed overall hematologic response rate (partial response, very good partial response, complete response) of isatuximab in relapsed/ refractory systemic light chain (AL) amyloidosis. Measured as rate of partial response or better.
  Partial response is defined as a dFLC decrease of ≥ 50%, but remaining > 4.0 mg/dL.
  Very good partial response is defined as the difference between involved and uninvolved FLCs [dFLC] < 4.0 mg/dL.
  Complete response is defined as laboratory values within the normal range free light chain (FLC) ratio (0.25 - 1.65) and negative serum and urine immunofixation.
Time Frame: From date of enrollment until progression or death due to any cause, whichever occurs first, assessed up to 4 years
Population: 35 participants who received treatment and are analyzable.
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Groups:
- Isatuximab: Patients receive isatuximab intravenously (IV) on days 1, 8, 15, and 22 of course 1 and on days 1 and 15 of subsequent courses. Treatment repeats every 28 days for 24 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Isatuximab
Number analyzed (Participants) | 35
percentage of paticipants | 77.1 [59.9 to 89.6]

2. Secondary Outcome: To Evaluate Toxicities in the Treatment of Relapsed/Refractory AL Amyloidosis With Isatuximab.
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: From date of enrollment until progression or death due to any cause, whichever occurs first, assessed up to 4 years
Population: Participants who completed at least one day of treatment.
Measure: Number; unit: Participants
Arm/Group | Isatuximab
Number analyzed (Participants) | 35
Participants
  Atrial fibrillation | 1
  Fatigue | 1
  Infections and infestations - Other, specify | 1
  Infusion related reaction | 1
  Lung infection | 2
  Lymphocyte count decreased | 3
  Pancreatitis | 1
  Pruritus | 1
  Skin infection | 1
  Syncope | 1

3. Secondary Outcome: Overall Survival (24 Month Estimate)
Description: Overall survival is measured from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact. While OS was assessed up to 4 years, 4 year estimates were not reached. We are reporting the 24 month estimate (how many participants reached survival time of at least 24 months).
Time Frame: From date of enrollment up to 2 years
Population: 35 eligible participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Isatuximab
Number analyzed (Participants) | 35
percent of participants | 85 [73 to 97]

4. Secondary Outcome: Duration of Response (24 Month Estimate)
Description: Duration of response is measure as time between hematologic response and hematologic progression.
  Hematologic progression is defined as 50% increase from nadir.
  While duration of response was assessed up to 4 years, 4 year estimates were not reached. We are reporting the 24 month estimate (how many participants achieved 24 month duration of response)
Time Frame: Up to 2 years
Population: 27 participants with response to study treatment
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Isatuximab
Number analyzed (Participants) | 27
Percent of Participants | 81 [67 to 96]

5. Secondary Outcome: Time to Hematologic Response
Description: To evaluate time to hematologic response. Partial response is defined as a dFLC decrease of ≥ 50%, but remaining > 4.0 mg/dL.
  Very good partial response is defined as the difference between involved and uninvolved FLCs [dFLC] < 4.0 mg/dL.
  Complete response is defined as laboratory values within the normal range free light chain (FLC) ratio (0.25 - 1.65) and negative serum and urine immunofixation.
Time Frame: From registration to time of confirmed hematologic progression
Population: Of the 35 analyzable participants, 27 achieved a response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Isatuximab
Number analyzed (Participants) | 27
Months | 1.1 [1 to 3]

6. Secondary Outcome: Progression-free Survival (24 Month Estimate)
Description: To evaluate progression-free survival (24 month estimate)
  Hematologic progression is defined as 50% increase from nadir, or from baseline (if there was no response) in any ONE OR MORE of the following:
  1. Serum M-protein: 50% increase in Serum M protein to a value greater than 0.5 g/dL.
  2. Urine M protein: 50% increase in Urine M protein to a value greater than 200 mg/day (a visible peak must be present)
  3. Free light chain increase of 50% to a value greater than 10 mg/dL
Time Frame: From registration to time of confirmed hematologic progression
Population: 35 participants were analyzable
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | Isatuximab
Number analyzed (Participants) | 35
percentage of paticipants | 74 [59 to 88]

ADVERSE EVENTS:
Time Frame: Up to 4 years after registration
Description: Participants who received protocol treatment and are eligible are included
Arm/Group | Isatuximab
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 15/35
Other Adverse Events (participants affected / at risk) | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Isatuximab (N=35)
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 1
Edema limbs (General disorders) | 1
Fever (General disorders) | 2
Bronchial infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Infections and infestations-Other (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Isatuximab (N=35)
Anemia (Blood and lymphatic system disorders) | 10
Blood and lymphatic system disorders-Other (Blood and lymphatic system disorders) | 2
Cardiac disorders-Other (Cardiac disorders) | 3
Heart failure (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 4
Sinus tachycardia (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 3
Cataract (Eye disorders) | 3
Dry eye (Eye disorders) | 3
Eye disorders-Other (Eye disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 18
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 4
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 10
Fever (General disorders) | 6
Gait disturbance (General disorders) | 2
General disorders and administration site conditio (General disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 5
Infections and infestations-Other (Infections and infestations) | 6
Lung infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 3
Upper respiratory infection (Infections and infestations) | 16
Urinary tract infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 6
Fall (Injury, poisoning and procedural complications) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 15
Injury, poisoning and procedural complications-Oth (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 2
Cardiac troponin I increased (Investigations) | 5
Cardiac troponin T increased (Investigations) | 2
Creatinine increased (Investigations) | 6
INR increased (Investigations) | 2
Investigations-Other (Investigations) | 5
Lymphocyte count decreased (Investigations) | 10
Weight gain (Investigations) | 2
Weight loss (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Muscle cramp (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal and connective tissue disorder - (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Neoplasms benign, malignant and unspecified (incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 8
Neuralgia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 6
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 7
Chronic kidney disease (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 2
Gynecomastia (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6
Respiratory, thoracic and mediastinal disorders-Ot (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 8
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03499808/Prot_SAP_002.pdf
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03499808/ICF_003.pdf